CLINICAL TRIAL: NCT04625413
Title: A Patient-centered Communication Tool (UR-GOAL) for Older Patients With Acute Myeloid Leukemia, Their Caregivers, and Their Oncologists
Acronym: UR-GOAL 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS20090
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Evaluate the usability and feasibility of a patient-centered communication tool (UR-GOAL)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Experimental Arm: single (Experimental): The UR-GOAL tool will incorporate conjoint analysis to elicit patient preferences as well as assessments of fitness and prognostic awareness.
  Interventions: Behavioral: Behavioral: UR-GOAL communication tool

INTERVENTIONS:
Behavioral: Behavioral: UR-GOAL communication tool — The UR-GOAL tool will incorporate conjoint analysis to elicit patient preferences as well as assessments of fitness and prognostic awarene

SUMMARY:
This is a pilot study to evaluate the usability and feasibility of a patient-centered communication tool (University of Rochester-Geriatric Oncology Assessment for acute myeloid Leukemia or UR-GOAL) among 15 older patients with AML, their caregivers, and oncologists.

DETAILED DESCRIPTION:
Older adults with AML and their caregivers may benefit from help and support in understanding their treatment options. This pilot study seeks to evaluate the usability and feasibility of the UR-GOAL communication tool. The UR-GOAL tool will incorporate conjoint analysis to elicit patient preferences as well as assessments of fitness and prognostic awareness.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Age ≥60 years (conventional definition of older age in AML)
* Newly diagnosed AML
* Considering treatment
* Able to provide informed consent
* English-speaking

Inclusion Criteria for Caregivers:

* Selected by the patient when asked if there is a "family member, partner, friend or caregiver [age 21 or older] with whom you discuss or who can be helpful in health-related matters;" patients who cannot identify such a person ("caregiver") can be eligible for the study. A caregiver need not be someone who lives with the patient or provides direct hands-on care. A caregiver can be any person who provides support (in any way) to the patient.
* Able to provide informed consent
* English-speaking

Inclusion Criteria for Oncologists:

* A practicing oncologist
* At least one of their patients are recruited to the study
* English-speaking

Exclusion Criteria: None

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-23 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete and final study protocol will be made publicly available through the University of Rochester Cancer Center Community Oncology Research Program Research Base Protocol and Data Sharing Committee. The full protocol and data will be made publicly available no later than the publication date of the study findings from the final dataset. The protocol will include a detailed description of the study population, hypotheses tested, measurement and assessment information, data definitions and codes, and the analysis plan utilized. We will be collecting identifying information. The final dataset will be stripped of identifiers prior to release for sharing. Published papers will be made available in portable document format.
Supporting Information: Study Protocol
Time Frame: The data will be available for 7 years from accrual of the first subject.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited older patients with AML, their caregivers, and oncologists from the University of Rochester Medical Center Wilmot Cancer Institute (WCI) and its affiliated oncology practices in upstate New York. Participants were recruited between October 2021 and March 2022.
Groups:
- Experimental: Experimental Arm: Single: The UR-GOAL tool will incorporate Best-Worst Scaling to elicit patient preferences as well as assessments of fitness and prognostic awareness.
  Behavioral: UR-GOAL communication tool: The UR-GOAL tool will incorporate Best-Worst Scaling to elicit patient preferences as well as assessments of fitness and prognostic awareness
Period: Overall Study
Arm/Group | Experimental: Experimental Arm: Single
Started | 15
Completed | 11
Not Completed | 4
Not completed — Hospice | 2
Not completed — Distress | 1
Not completed — Not feeling well | 1

BASELINE CHARACTERISTICS:
Population: Older adults aged 60 and over
Arm/Group | Experimental: Experimental Arm: Single
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Feasibility (Recruitment Rates)
Description: Percentage of patients who consented to the study ultimately completed the study intervention and post-intervention assessment
Time Frame: Four weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Experimental Arm: Single
Number analyzed (Participants) | 15
Participants | 11

2. Primary Outcome: Usefulness
Description: Usefulness was assessed using the Preparation for Decision Making Scale (mean score range from 1 to 5, and higher scores indicate greater usefulness)
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Experimental Arm: Single
Number analyzed (Participants) | 11
score on a scale | 3.8 (0.7)

3. Secondary Outcome: Pre-post Changes in the Following Outcomes:Perceived Efficacy in Patient-Physician Interactions (PEPPI)
Description: A valid and reliable assessment of perceived self-efficacy of older patients interacting with physicians; score on 5-item scale, ranging 5-25; higher score corresponds to greater perceived efficacy. Pre-post changes from baseline to four weeks.
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Experimental Arm: Single
Number analyzed (Participants) | 11
score on a scale | 1.5 (3.0)

4. Secondary Outcome: Pre-post Changes in the Following Outcomes: General Anxiety Disorder-7
Description: A 7-item screening tool for anxiety; ranging 7-21; higher score corresponds to greater anxiety symptoms. Pre-post changes from baseline to four weeks.
Time Frame: Four weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental: Experimental Arm: Single: The UR-GOAL tool will incorporate Best-Worst Scaling to elicit patient preferences as well as assessments of fitness and prognostic awareness.
  Behavioral: UR-GOAL communication tool: The UR-GOAL tool will incorporate est-Worst Scaling to elicit patient preferences as well as assessments of fitness and prognostic awarene
Arm/Group | Experimental: Experimental Arm: Single
Number analyzed (Participants) | 11
score on a scale | -1.6 (5.4)

5. Secondary Outcome: Pre-post Changes in the Following Outcomes: Geriatric Depression Scale-15
Description: A 15-item valid and reliable screening tool for depression in older adults. This will be used for patients; ranging 0-15; higher score corresponds to greater depressive symptoms. Pre-post changes from baseline to four weeks.
Time Frame: Four Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental: Experimental Arm: Single: The UR-GOAL tool will incorporate Best-Worst Scaling to elicit patient preferences as well as assessments of fitness and prognostic awareness.
  Behavioral: UR-GOAL communication tool: The UR-GOAL tool will incorporate Best-Worst Scaling to elicit patient preferences as well as assessments of fitness and prognostic awarene
Arm/Group | Experimental: Experimental Arm: Single
Number analyzed (Participants) | 11
score on a scale | 0.2 (2.1)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Experimental: Experimental Arm: Single
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT04625413/Prot_SAP_000.pdf